CLINICAL TRIAL: NCT02310113
Title: Red Blood Cell Transfusion and Skeletal Muscle Tissue Oxygenation in Anaemic Haematologic Outpatients
Brief Title: Transfusion and Skeletal Muscle Tissue Oxygenation
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Podbregar Matej, Prof., University Medical Centre Ljubljana
Other Study IDs: Anemia_NIRS
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Anemia
Keywords: NIRS; transfusion; RBC
MeSH Terms: conditions — Anemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hematologic outpatients: Chronic anaemic outpatients who are planed to get transfusion RBC
  Interventions: Other: NIRS

INTERVENTIONS:
Other: NIRS — Measurment of skeletal muscle oxygenation by near-infrared spectroscopy
  Other Names: near infrared spectroscopy

SUMMARY:
The aim of the present study was to re-challenge the current data that anaemia in chronically anaemic haematology patients is not associated with low skeletal muscle StO2, and that the age of RBCs does not influence tissue responses. The investigators investigated these aspects using improved technology NIRS devices, for deeper tissue penetration and removal of the superficial signal from the skin.

DETAILED DESCRIPTION:
Anaemia is state of decreased blood oxygen carrying capacity . Acute anaemia is associated with increased tissue oxygen extraction . On the other hand, with chronic anaemia human body has time to at least partially adapt to decreased blood oxygen carrying capacity , .

Near-infrared spectroscopy (NIRS) is non-invasive method to assess tissue oxygenation (StO2) and estimate tissue haemoglobin (THb) levels . The investigators have studied skeletal muscle StO2 in critically ill patients with preserved oxygen (i.e., cardiogenic shock) and with impaired oxygen extraction (i.e., septic shock) , , . In addition to measuring resting StO2, the investigators performed vascular occlusion tests to stop arterial blood flow, to estimate oxygen consumption, and at the end of the occlusion, it was also possible to estimate vascular reactivity and maximal reperfusion capability .

Under acute blood loss in trauma patients, the skeletal muscle StO2 measured by NIRS correlates with blood haemoglobin (Hb) and delivery of oxygen, and can easily detect latent stage of haemorrhagic shock . Unexpectedly, chronically anaemic haematology patients with preserved oxygen extraction capability did not show low skeletal StO2 and THb index despite their severe anaemia, which is what would be predicted from normal physiological responses .

It is known that there are structural and functional changes to RBCs during storage. Recent study detected deleterious effects of RBC storage on microvascular responses to transfusion in stable anaemic trauma patients .

The aim of the present study was to re-challenge the current data that anaemia in chronically anaemic haematology patients is not associated with low skeletal muscle StO2, and that the age of RBCs does not influence tissue responses. The investigators investigated these aspects using improved technology NIRS devices, for deeper tissue penetration and removal of the superficial signal from the skin.

ELIGIBILITY:
Inclusion Criteria:

* chronic haematologic patients

Exclusion Criteria:

* pregnancy
* rejection to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematologic anaemic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
basal Sto2 | 1 hour
  change of basal Sto2 of skeletal muscle after RBC transfusion

SECONDARY OUTCOMES:
vascular occlusion testing | 5 minutes
  measuring of dynamic tissue oxygenaion

CONTACTS AND LOCATIONS:
Overall Officials: matej podbregar, MD PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- Clinical Center Ljubljana, Ljubljana, Slovenia